CLINICAL TRIAL: NCT01089283
Title: I123 DAT-SCAN and PET-CT FDG to Assess Brain Function of Parkinson Patients With Different Genetic Characteristic
Brief Title: Ioflupane I123 (DaTSCAN) and Positron Emission Tomography-computed Tomography Fludeoxyglucose (PET-CT FDG) to Assess Brain Function of Parkinson Patients With Different Genetic Characteristics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD. Head, Dept of Nuclear Medicine, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-EES-087-CTIL
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson Disease
Keywords: parkinson; fdg pet-ct; i123 dat scan; LRRK2; GBA; parkinson patients with known genetic characteristic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- LRRK2 mutation: Parkinson patients that carry mutation on LRRK2 gene
- GBA mutation: Parkinson patients that carry mutation on GBA gene
- no mutation: Parkinson patients that don't carry mutation on LRRK2 or GBA genes
- healthy: Healthy volunteers

SUMMARY:
Parkinson disease is one of the most common neurodegenerative illnesses. The disease is characterized by decrease in dopamine levels and decrease in the number of dopaminergic neurons and dopamine receptors. There are gene mutations that increase the risk for the disease. Two of those mutations are on the LRRK2 gene and on GBA gene. It is yet unknown if there is a difference between the metabolic brain function of Parkinson patients that carry one of the two mutations to Parkinson patients with no known mutation.

Participants: diagnosed Parkinson patients that carry a gene mutation in either LRRK2 or GBA genes, Parkinson patients with no known mutation and healthy volunteers as a control group.

The participants will go through both examinations DAT SCAN and PET CT SCAN at the Tel Aviv Sourasky Medical Center Nuclear Medicine Institute.

The examination results will be given to the participants by a doctor from the neurology department.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Parkinson patients with known genetic characteristics

Exclusion Criteria:

* patients unable to understand and sign an informed consent
* minors
* patients in medical condition that does not allow them to stay still during the examination

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed parkinson patients ages: 40-80
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, MD, PhD, Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Volkow ND, Ding YS, Fowler JS, Wang GJ, Logan J, Gatley SJ, Hitzemann R, Smith G, Fields SD, Gur R. Dopamine transporters decrease with age. J Nucl Med. 1996 Apr;37(4):554-9. PMID 8691238
- [Background] Huang Y, Cheung L, Rowe D, Halliday G. Genetic contributions to Parkinson's disease. Brain Res Brain Res Rev. 2004 Aug;46(1):44-70. doi: 10.1016/j.brainresrev.2004.04.007. PMID 15297154
- [Background] Vila M, Przedborski S. Genetic clues to the pathogenesis of Parkinson's disease. Nat Med. 2004 Jul;10 Suppl:S58-62. doi: 10.1038/nm1068. PMID 15272270
- [Background] von Bohlen und Halbach O, Schober A, Krieglstein K. Genes, proteins, and neurotoxins involved in Parkinson's disease. Prog Neurobiol. 2004 Jun;73(3):151-77. doi: 10.1016/j.pneurobio.2004.05.002. PMID 15236834
- [Background] Farrer M, Stone J, Mata IF, Lincoln S, Kachergus J, Hulihan M, Strain KJ, Maraganore DM. LRRK2 mutations in Parkinson disease. Neurology. 2005 Sep 13;65(5):738-40. doi: 10.1212/01.wnl.0000169023.51764.b0. PMID 16157908
- [Background] Orr-Urtreger A, Shifrin C, Rozovski U, Rosner S, Bercovich D, Gurevich T, Yagev-More H, Bar-Shira A, Giladi N. The LRRK2 G2019S mutation in Ashkenazi Jews with Parkinson disease: is there a gender effect? Neurology. 2007 Oct 16;69(16):1595-602. doi: 10.1212/01.wnl.0000277637.33328.d8. PMID 17938369
- [Background] Herholz K, Heiss WD. Positron emission tomography in clinical neurology. Mol Imaging Biol. 2004 Jul-Aug;6(4):239-69. doi: 10.1016/j.mibio.2004.05.002. PMID 15262239
- [Background] Pavese N, Brooks DJ. Imaging neurodegeneration in Parkinson's disease. Biochim Biophys Acta. 2009 Jul;1792(7):722-9. doi: 10.1016/j.bbadis.2008.10.003. Epub 2008 Oct 17. PMID 18992326
- [Background] Ozelius LJ, Senthil G, Saunders-Pullman R, Ohmann E, Deligtisch A, Tagliati M, Hunt AL, Klein C, Henick B, Hailpern SM, Lipton RB, Soto-Valencia J, Risch N, Bressman SB. LRRK2 G2019S as a cause of Parkinson's disease in Ashkenazi Jews. N Engl J Med. 2006 Jan 26;354(4):424-5. doi: 10.1056/NEJMc055509. No abstract available. PMID 16436782
- [Background] Thaler A, Ash E, Gan-Or Z, Orr-Urtreger A, Giladi N. The LRRK2 G2019S mutation as the cause of Parkinson's disease in Ashkenazi Jews. J Neural Transm (Vienna). 2009 Nov;116(11):1473-82. doi: 10.1007/s00702-009-0303-0. PMID 19756366
- [Background] Hassin-Baer S, Laitman Y, Azizi E, Molchadski I, Galore-Haskel G, Barak F, Cohen OS, Friedman E. The leucine rich repeat kinase 2 (LRRK2) G2019S substitution mutation. Association with Parkinson disease, malignant melanoma and prevalence in ethnic groups in Israel. J Neurol. 2009 Mar;256(3):483-7. doi: 10.1007/s00415-009-0117-x. Epub 2009 Mar 24. PMID 19412725
- [Background] Gan-Or Z, Giladi N, Rozovski U, Shifrin C, Rosner S, Gurevich T, Bar-Shira A, Orr-Urtreger A. Genotype-phenotype correlations between GBA mutations and Parkinson disease risk and onset. Neurology. 2008 Jun 10;70(24):2277-83. doi: 10.1212/01.wnl.0000304039.11891.29. Epub 2008 Apr 23. PMID 18434642
- [Derived] Artzi M, Even-Sapir E, Lerman Shacham H, Thaler A, Urterger AO, Bressman S, Marder K, Hendler T, Giladi N, Ben Bashat D, Mirelman A. DaT-SPECT assessment depicts dopamine depletion among asymptomatic G2019S LRRK2 mutation carriers. PLoS One. 2017 Apr 13;12(4):e0175424. doi: 10.1371/journal.pone.0175424. eCollection 2017. PMID 28406934